CLINICAL TRIAL: NCT06243237
Title: Efficacy of Acupuncture in Patients With Acute Intracranial Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202201836A3
Record Dates: First submitted 2023-12-19; First posted 2024-02-06 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-12

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group(acupuncture group) (Experimental): After blind random allocation, investigators applied acupuncture on patient with acute intracranial hemorrhage.
  Interventions: Procedure: Acupuncture
- Control group(sham acupuncture group (superficial acupuncture)) (Placebo Comparator): After blind random allocation, investigators applied superficial acupuncture on patient with acute intracranial hemorrhage.
  Interventions: Procedure: Sham Acupuncture(Superficial Acupuncture)

INTERVENTIONS:
Procedure: Acupuncture — Applied acupuncture on specific acupoints in patient with acute intracranial hemorrhage.
  Arms: Intervention group(acupuncture group)
Procedure: Sham Acupuncture(Superficial Acupuncture) — Applied superficial acupuncture on specific acupoints in patient with acute intracranial hemorrhage.
  Arms: Control group(sham acupuncture group (superficial acupuncture))

SUMMARY:
Investigators propose a research design protocol to evaluate the efficacy of acupuncture in improving function recovery after acute intracranial hemorrhage.

DETAILED DESCRIPTION:
Stroke is a major cause of death and disability. According to the Ministry of Health and Welfare in Taiwan, stroke accounted for 6.8% of all deaths and was the 4th leading cause of death in Taiwan in 2020. Stroke can be divided into acute, subacute, and chronic stages, and the initial severity of stroke affects recovery from sequelae. Therefore, how to effectively improve the sequelae and accelerate the recovery of patients through early interventions is an important issue. This study aimed to investigate the effect of early acupuncture treatment in the acute stage of hemorrhagic stroke. Subjects will be divided into two main groups by random assignment. The intervention group will be treated with traditional acupuncture, while the control group will be treated with pseudo-acupuncture(superficial acupuncture). The treatment frequency was 3 times a week for at least one week. Consciousness, neurological status and disability status were assessed before treatment, at the end of the first week, the second week and the third week, and biomarker were examined before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemorrhagic stroke by a specialist
* Age over 20 years and below 85 years
* GCS between 5-13

Exclusion Criteria:

* Intracranial hemorrhage resulted from vascular anomalies
* Pregnant patients
* Intracranial tumor related hemorrhage
* Other diseases that can cause neurological deficits, such as old cerebrovascular disease, poliomyelitis, cerebral palsy, spinal cord injury
* Organ damage or terminal illness (heart or kidney failure or malignancy)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | 3 weeks and follow-up for one year
  The Barthel Index is a scale used to measure performance in activities of daily living (ADL). The total score can range from 0 (complete dependence) to 100 (complete independence), providing a quantitative measure of an individual's functional independence.
Muscle Power | 3 weeks and follow-up for one year
  Muscle power is often assessed using a grading system. The most common is the Medical Research Council (MRC) Scale, which grades muscle strength on a scale from 0 to 5 and the lower scores mean the worse outcome.
The Modified Rankin Scale | 3 weeks and follow-up for one year
  The Modified Rankin Score (mRS) is a scale with scores ranging from 0 to 6, the higher scores mean the worse outcome.
National Institute of Health Stroke Scale | 3 weeks and follow-up for one year
  The total NIHSS score can range from 0 to 42, where a score of 0 means no stroke symptoms, and a higher score indicates a more severe stroke.
Glasgow Coma Scale(GCS) | 3 weeks and follow-up for one year
  The Glasgow Coma Scale(GCS) is a clinical scale used to reliably measure a person's level of consciousness. The total score can range from 3 to 15, and the lower scores mean the worse outcome.
Karnofsky Performance Scale | 3 weeks and follow-up for one year
  The Karnofsky Performance Score (KPS) ranking runs from 100 to 0, where 100 is "perfect" health and 0 is death.

SECONDARY OUTCOMES:
Pulse analysis system (PPAS-96)(Sphygmography) | 3 weeks and follow-up for one year
  Pulse analysis system (PPAS-96) can realize the digitization of pulse wave graphics, establish a pulse wave database (scale unit: Hertz, Hz).
Completed blood count (CBC) | 3 weeks and follow-up for one year
  Measuring the amounts of red blood cells (RBC, million/μL), white blood cells (WBC, 1000/μL), platelets (Plt, 1000/μL), along with the hemoglobin (Hb, g/dL) and hematocrit (Hct, %) values via automated hematology analyzer.
White blood cells differential count | 3 weeks and follow-up for one year
  Calculating the percentage of each type of white blood cell (WBC): Segment(%), Band(%), Lymphocyte(%), Monocyte(%), Eosinophil(%), Basophil(%)
C reactive protein (CRP) | 3 weeks and follow-up for one year
  Measuring the level of C reactive protein in blood. (CRP, mg/L)
Albumin | 3 weeks and follow-up for one year
  Measuring the level of albumin in blood. (Alb, g/dL)
Blood urea nitrogen (BUN) | 3 weeks and follow-up for one year
  Measuring the level of blood urea nitrogen. (BUN, mg/dL)
Creatinine | 3 weeks and follow-up for one year
  Measuring the level of creatinine in blood. (Crea, mg/dL)
Sodium | 3 weeks and follow-up for one year
  Measuring the level of sodium in blood. (Na, milliequivalent (mEq)/L)
Potassium | 3 weeks and follow-up for one year
  Measuring the level of potassium in blood. (K, milliequivalent (mEq)/L)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ru Ko, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang-Gung Memorial Hospital, Keelung, Taiwan